CLINICAL TRIAL: NCT04580992
Title: Defining the Electrocardiographic Effect of Propofol on the Ajmaline Provocation Drug Challenge: A Prospective Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: APA Brugada study
Record Dates: First submitted 2020-10-01; First posted 2020-10-09 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-09

CONDITIONS: Brugada Syndrome; Channelopathies; Ventricular Fibrillation; Cardiac Death
MeSH Terms: conditions — Brugada Syndrome; Channelopathies; Ventricular Fibrillation; Death | interventions — Ajmaline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ajmaline group
  Interventions: Drug: Ajmaline

INTERVENTIONS:
Drug: Ajmaline — Ajmaline administration

SUMMARY:
Background: Brugada Syndrome is an inherited channelopathy associated with risk of ventricular fibrillation and sudden cardiac death in a structurally normal heart. The diagnosis is based on the characteristic electrocardiographic pattern (coved type STsegment elevation, 2mm followed by a negative T-wave in one or more of the right precordial leads V1 to V2), noted spontaneously or upon administration of a sodiumchannel blocker, such as Ajmaline.

The majority of adults screened for Brugada Syndrome, undergo the Ajmaline provocation-test awake. Ajmaline is therefore injected continuously, with incremental steps through an intravenous placed catheter, according to cardiological protocols. In a subpopulation of anxious adults, or when another electrophysiological procedure is required at the same time, sedation or general anaesthesia is provided. Similarly, in the paediatric population, it is common practice to perform the challenge test under sedation.

Based on the sodium channel blocking properties of propofol, it is not unthinkable that anaesthetic agents might interact with the pharmacodynamic or pharmacokinetic effects of Ajmaline on the myocardial sodium channels. Existence of such interaction would implicate altered diagnostic value of the Ajmaline-provocation-test for patients that undergo the challenge under general anaesthesia.

Objective: The goal of this study is to evaluate if the Ajmaline-provocation-test results in altered electrocardiographic effects when performed under general anaesthesia with propofol.

Study-design: A prospective observational study.

Study population: Patients are eligible for inclusion if they have been diagnosed with Brugada Syndrome, are American Society of Anaesthesiologists (ASA) 2 - 4, older than 18 years and are scheduled for epicardial ablation. Exclusion criteria are known allergy for propofol, a body mass index (BMI) above 35 for female and 42 for male patients, obstetric patients, critical illness, conditions that exclude continuous propofol infusion due to higher risk for propofol infusion syndrome (PRIS), such as mitochondrial disease, fatty acid oxidation disorder, co-enzyme Q deficiency and any other condition that renders the patient unfit for elective surgery.

Intervention: This study is prospective, observational.

Main study parameters/endpoints: The primary endpoints are changes in the ST-, Jp-, QRS-, T(p-e)-segments and T(p-e)/QT -ratio changes during steady-state anaesthesia. The secondary endpoint is the occurrence of de novo arrhythmias.

Nature and extent of the burden and risks associated with participation: This is an observational study; therefore, the risks associated are no other than those associated with the intervention itself. No additional blood-samples, tests or consults are necessitated during participation; therefore, no extra burden is associated.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 year
* ASA 2, 3, 4
* Epicardial ablation indicated by cardiologist
* Written informed consent

Exclusion Criteria:

* A known allergy to propofol
* BMI>35 for female patients
* BMI > 42 for male patients
* Obstetric anaesthesia
* Critical Illness
* Mitochondrial disease
* Fatty acid oxidation disorder
* Co-enzyme Q deficiency
* Any condition that renders the patient unfit for elective surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are eligible for inclusion upon the age of 18, diagnosed with Brugada Syndrome and when epicardial ablation was indicated as treatment. In this study, we would like to include at least twenty-five patients.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
ST-, QRS-, Jp-, QT-, QTcB-, QTcFr- and JT-interval | during the intervention/procedure/surgery
  Ventricular Arrhythmogenesis

SECONDARY OUTCOMES:
Malignant arrhythmias | intra- or postoperatively (up to 24hours upon discharge from the post anaesthetic care unit)
  Previously not-known or non-existing ventricular or supraventricular arrhythmias resulting in compromising hemodynamic instability detrimentally affecting cardiac output and requiring advanced cardiac life treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussels, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided